CLINICAL TRIAL: NCT02359773
Title: Two Cohort, Pilot Study, to Identify Magnetocardiogram Characteristics That Can be Used to Classify Non Ischemic Chest Pain Patients and Myocardial Infarction Patients.
Brief Title: Magnetocardiography as a Tool for Patients Presenting With Chest Pain - Pilot Study
Status: Completed | Type: Observational
Sponsor: Quantum Imaging Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: QI CIP 001 Rev 001
Record Dates: First submitted 2015-01-12; First posted 2015-02-10 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-02

CONDITIONS: Chest Pain
Keywords: Magnetocardiography; Myocardial Infarction; Non-ischaemic chest pain
MeSH Terms: conditions — Chest Pain; Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group 1 - Non ischemic chest pain: No coronary artery disease (CAD) as confirmed by myoview, MRI or stress echo. Subjects will receive one MCG scan (intervention) using the QI Model 1.0 Magentocardiogram. This will be in addition to their current care and it will not be used to support clinical decision making.
- Group 2 - Myocardial infarction: Myocardial infarction confirmed by a troponin test (>50ng/l) 12 hours after the onset of chest pain. Subjects will receive one MCG scan (intervention) using the QI Model 1.0 Magentocardiogram. This will be in addition to their current care and it will not be used to support clinical decision making.

SUMMARY:
The purpose of this pilot research study is to identify the characteristics of magnetocardiograms that correlate with a non ischemic chest pain status and a myocardial infarction patient status. The study uses a non SQUID magnetocardiogram device.

DETAILED DESCRIPTION:
Magnetocardiography (MCG) is a passive, non-contact technique to measure the electromagnetic activity of the heart.

Heart muscle is controlled by electrical impulses that initiate contraction of the myocardium to pump blood around the body. A wave of depolarisation and repolarisation helps to coordinate the heart's activity which is usually measured using an electrocardiogram (ECG) which reflects the surface electrical manifestation of myocardial depolarisation and repolarisation

For every electrical signal there is a corresponding magnetic field, as defined by Faraday's law of induction, and it is this magnetic field that MCG measures.

There are two key advantages of looking at the magnetic field rather than the electrical signal. (1) The signal is not attenuated as it passes through the body, so information is not lost and (2) changes in the action potential (for example those caused by ischemia) are 'magnified' in the magnetic field so are easier to detect by sensors that are not in direct contact with the body.

SQUID MCG has been used widely in cardiology research, and previous clinical studies have shown that the technology has potential for the analysis of patients with coronary artery disease.

The aim of this pilot study is to identify characteristics of MCG that differentiate patients with non-ischaemic chest pain from those with a myocardial infarction.

.

ELIGIBILITY:
Inclusion Criteria:

Non ischemic chest pain subject inclusion criteria

* Subjects will be males or females over the age of 18.
* Subjects will have experienced chest pain within the last 8 weeks and have been subsequently referred to the rapid access chest pain clinic (RACPC).
* Subjects will have no coronary artery disease/ischemia as demonstrated by one of the following: MRI, myoview or stress echo within no less than 4 weeks prior to the magnetocardiogram (MCG) scan.
* Subjects will have given written informed consent to participate in the study.

Myocardial Infarction subject inclusion criteria

* Subjects will be males or females over the age of 18.
* Subjects will have experienced chest pain and have been admitted to the cardiology unit.
* Subjects will have an abnormal level of Troponin (≥50ng/l) taken at 12 hours following the onset of chest pain.
* Subjects will be suitable to have an MCG scan taken within 48 hours of the onset of chest pain and prior to coronary angioplasty or any other surgical intervention.
* Subjects will have given written informed consent to participate in the study.

Exclusion Criteria:

Non ischemic chest pain subject exclusion criteria

* Subjects with symptoms suggestive of acute coronary syndrome that require further investigation.
* Subjects who had an abnormal level of Troponin (≥50ng/l) - as determined by a test performed prior to referral to the RACPC.
* Subjects who have a pacemaker or internal cardiac defibrillator.
* Subjects with an active implantable device.
* Subjects with ferrous implants in the torso including wires or ferrous stents.
* Subjects who are pregnant.
* Subjects who are unable to lie in a supine position.
* Subjects with any comorbidity that prevents them being scanned.

Myocardial Infarction subject exclusion criteria

* Subjects who have had a STEMI.
* Patients with haemodynamic instability (dysrhythmia or hypotension).
* Subjects who have had a revascularisation technique performed prior to an MCG scan.
* Subjects who have a pacemaker or internal cardiac defibrillator.
* Subjects with ferrous implants in the torso including wires or ferrous stents.
* Subjects with an active implantable device.
* Subjects who are pregnant.
* Subjects who are unable to lie in a supine position.
* Subjects with any comorbidity that prevents them being scanned.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting in Accident and Emergency Department with chest pain of presumed ischemic origin
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2015-02; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Magnetocardiogram Characteristics in patients with chest pain | 1 hour
  Quantitative comparison of magnetocardiogram characteristics of non ischaemic chest pain patients compared to those with an acute myocardial infarction

SECONDARY OUTCOMES:
Device Safety | At time of scan for all patiients (Varies)
  Any adverse effects, adverse device effects, Unanticipated serious device effects

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kearney, MBChB FRCP, Principal Investigator — Leeds Teaching Hospitals NHS Trust
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom